CLINICAL TRIAL: NCT01103011
Title: A Phase I, Single Center, Blinded, Controlled Study Evaluating Safety, Tolerability and Pharmacokinetic Profile of Levodopa Following Repeated Administration of Oral Levodopa/Carbidopa and Continuously Delivered ND0611
Brief Title: Safety, Tolerability and Pharmacokinetic Profile of Levodopa Administered With Continuous Administration of ND0611
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroDerm Ltd. (Industry)
Responsible Party: Sheila Oren MD, VP Clinical and Regulatory Affairs, Neuroderm, ltd.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ND0611/001
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- ND0611 dose 1, ND0611 dose 2, placebo (Experimental)
  Interventions: Drug: ND0611

INTERVENTIONS:
Drug: ND0611 — Continuous delivery of ND0611
Drug: ND0611 — Solution of ND0611 delivered continuously

SUMMARY:
The study hypothesis is that continuous ND0611 increases the bioavailability of levodopa and therefore the levodopa area-under-the-concentration-curve values, half-life, and trough concentrations The study will help determining the safety and tolerability of ND0611 and determine the pharmacokinetic profile of levodopa following multiple oral dosing of levodopa/carbidopa (LD/CD) and continuous delivery of ND0611

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian males between 18 and 50 years (inclusive) of age
* Normal body weight
* Subjects with negative urinary drugs of abuse, HIV, Hepatitis B or Hepatitis C serology tests
* Subjects must be able to adhere to the protocol requirements
* Subjects must provide written informed consent to participate in the study.
* Haemoglobin level >12.5 mg /dl

Exclusion Criteria:

* History of significant psychiatric disorder, neurological diseases or sleep disorders
* History of significant systemic diseases, by medical history or tests performed during screening examinations
* Clinically significant laboratory tests at screening
* History of drug or alcohol abuse.
* Allergy to levodopa, carbidopa or any inactive component of the test formulation.
* Subjects with dark skin
* Subjects with skin diseases or neoplasms
* Subjects with narrow-angle glaucoma
* Subjects with significant allergic response to other drugs.
* Subject with known atopic disorders
* Known allergy or hypersensitivity to adhesive tapes.
* Use of any prescription or over-the-counter (OTC) medications
* Subjects who donated blood or received blood, in the last 3 months
* Participation in another clinical trial in the last 30 days
* Subjects which do not have the ability to communicate well or will not adhere to the protocol procedures

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability
  Safety and tolerability:
  * Adverse event reporting
  * Discontinuation of the treatment due to adverse event

SECONDARY OUTCOMES:
Pharmacokinetics
  Pharmacokinetic profile of plasma LD and CD:
  * Primary endpoint: t½
  * Secondary endpoints: through levels, Cmax, Tmax, AUC

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel